CLINICAL TRIAL: NCT07305194
Title: Study of Atrial High-Rate Episode Burden in Patients Undergoing Concurrent Bachmann Bundle Area Pacing and Left Bundle Branch Pacing , Compared With Either Left Bundle Branch Pacing or Conventional Right Ventricular Pacing.
Brief Title: Study of AHRE Burden in Patients Undergoing Bachmann Bundle Area Pacing and Left Bundle Branch Pacing.
Acronym: AHRE-BLAST
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Georgios Leventopoulos, Assistant Professor of Cardiology - Electrophysiology Patras University Hospital, Greece, University Hospital of Patras
Other Study IDs: UHP-LBBP-BBP-AHRE-2025
Record Dates: First submitted 2025-11-18; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Atrial Arrhythmia; Atrial Fibrillation (AF); Pacemaker Implantation; Left Bundle Branch Pacing; Conduction System Pacing
Keywords: Atrial High-Rate Episodes (AHRE); Subclinical Atrial Fibrillation; Bachmann Bundle Area Pacing (BBAP); Left Bundle Branch Pacing (LBBP); Physiological Pacing; Interatrial Conduction; Atrial Synchrony; P-wave Duration; Atrial Electromechanical Remodeling; Atrial Strain; Left Atrial Reservoir Strain; Inter-atrial Conduction Delay (IACD); Speckle Tracking Echocardiography; Left Atrial Volume Index (LAVI); Atrial Arrhythmias; Device-Detected AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Concurrent BBAP + LBBP (total physiological pacing)
- RAA pacing + LBBP
- Conventional pacing (RAA + RV pacing)

SUMMARY:
This prospective observational study evaluates the burden of Atrial High-Rate Episodes (AHRE) in patients without a prior history of atrial fibrillation who undergo concurrent Bachmann Bundle Area Pacing (BBAP) and Left Bundle Branch Pacing (LBBP). Physiological pacing at these sites aims to improve interatrial conduction and reduce the risk of atrial arrhythmias.

The study includes a comparative assessment across three patient groups:

1. BBAP + LBBP (physiological pacing group)
2. Right Atrial Appendage (RAA) pacing + LBBP
3. Conventional pacing - RAA and Right Ventricular (RV) pacing AHRE burden will be quantified via device diagnostics and remote monitoring at 3, 12 and 24 months post-implantation. Episodes will be classified by duration (0-6 min, 6-24 h, >24 h), differentiating subclinical AHRE from clinically documented AF.

Secondary analyses include electrocardiographic changes (P-wave indices), the need for antiarrhythmic therapy, and comprehensive echocardiographic evaluation of atrial function (e.g., LA strain, conduction delays, LAVI).

The study aims to determine whether physiological pacing (BBAP + LBBP) provides superior protection against AHRE development compared with RAA + LBBP and conventional pacing strategies.

DETAILED DESCRIPTION:
Atrial high-rate episodes (AHRE) detected by cardiac implantable devices are associated with an increased risk of developing atrial fibrillation (AF), stroke, and atrial remodeling. Traditional right atrial and right ventricular pacing may alter atrial activation patterns, potentially promoting electrical and structural changes that predispose to atrial arrhythmias.

Physiologic pacing strategies targeting the Bachmann bundle region and the left bundle branch have emerged as alternatives designed to preserve normal conduction pathways. Bachmann Bundle Area Pacing (BBAP) facilitates more synchronous biatrial activation, while Left Bundle Branch Pacing (LBBP) results in near-physiologic ventricular activation. Both methods may reduce conduction delays and improve atrial and ventricular electromechanical function.

This prospective observational study examines whether physiologic atrial and ventricular pacing reduces the burden of device-detected AHRE compared with commonly used pacing configurations. Three groups are evaluated: (1) BBAP combined with LBBP, (2) right atrial appendage pacing combined with LBBP, and (3) conventional right atrial and right ventricular pacing. All enrolled participants have a clinical indication for permanent pacing and no prior diagnosis of AF.

AHRE burden will be assessed through routine device diagnostics and remote monitoring over a 24-month follow-up. Electrocardiographic and echocardiographic data will also be collected to explore relationships between conduction patterns, atrial function, and arrhythmia occurrence. The study aims to clarify whether preserving physiologic conduction pathways influences long-term AHRE burden and may contribute to AF prevention in paced patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with a clear indication for permanent pacing, according to ESC guidelines [15] for the management of conduction disturbances (e.g. symptomatic bradycardia, complete atrioventricular block, sinus node dysfunction).
* Sinus rhythm at the time of implantation, with no documented episodes of atrial fibrillation prior to implantation, either in the medical history or in previous recordings (ECG, Holter, telemetry).
* Ability to be followed up for at least 24 months after implantation.
* Provision of written informed consent to participate in the study.

Exclusion Criteria:

* History of atrial fibrillation prior to implantation, either permanent or paroxysmal, documented on ECG, Holter, or telemetry.
* Prior pharmacological or interventional treatment for AF (e.g. antiarrhythmic drugs, catheter ablation).
* Inability to comply with long-term follow-up or non-adherence to follow-up visits.
* Contraindications to pacemaker lead placement at the selected sites.
* Participation in another study that could influence the results.
* Previous device implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) with a clear indication for permanent pacing, according to ESC guidelines [15] for the management of conduction disturbances (e.g. symptomatic bradycardia, complete atrioventricular block, sinus node dysfunction).
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-05 (Estimated); Study Completion 2028-04-14 (Estimated)

PRIMARY OUTCOMES:
AHRE burden | 24 months
  PRIMARY OUTCOME MEASURE Unit of measure : percent (%) AHRE Burden (% of monitored time) Percentage of total monitored time spent in device-detected atrial high-rate episodes (AHRE), as defined by manufacturer diagnostic criteria

SECONDARY OUTCOMES:
Number of AHRE episodes (0-6 minutes ) | 24 months
  Device-detected AHRE episodes lasting 0-6 minutes. Unit of measure: Number of episodes
Number of AHRE Episodes (6 minutes-24 hours) | 24 months
  Device-detected AHRE episodes lasting 6 minutes to 24 hours. Unit of Measure: Number of episodes
Number of AHRE Episodes (>24 hours) | 24 months
  Device-detected AHRE episodes lasting more than 24 hours. Unit of measure: Number of episodes
Incidence of Clinically Documented Atrial Fibrillation | 24 months
  Clinically confirmed AF episodes identified via ECG or rhythm strip. Unit of measure : number of events
Maximum P-Wave Duration | Baseline, 24 months
  Maximum P-wave duration measured on 12-lead ECG Unit of measure : Milliseconds (ms)
P - wave axis | Baseline, 24 months
  Frontal plane P-wave axis measured on 12-lead ECG Unit of Measure: Degrees
Initiation or Modification of Antiarrhythmic Therapy | Baseline, 24 months
  Number of participants requiring initiation or change in antiarrhythmic. Unit of Measure: Number of participants

CONTACTS AND LOCATIONS:
Locations (1):
- University General Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Michael Glikson et al., 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: Developed by the Task Force on cardiac pacing and cardiac resynchronization therapy of the European Society of Cardiology (ESC) With the special contribution of the European Heart Rhythm Association (EHRA), European Heart Journal, Volume 42, Issue 35, 14 September 2021, Pages 3427-3520, https://doi.org/10.1093/eurheartj/ehab364.
- [Result] Glotzer TV, Hellkamp AS, Zimmerman J, Sweeney MO, Yee R, Marinchak R, Cook J, Paraschos A, Love J, Radoslovich G, Lee KL, Lamas GA; MOST Investigators. Atrial high rate episodes detected by pacemaker diagnostics predict death and stroke: report of the Atrial Diagnostics Ancillary Study of the MOde Selection Trial (MOST). Circulation. 2003 Apr 1;107(12):1614-9. doi: 10.1161/01.CIR.0000057981.70380.45. Epub 2003 Mar 24. PMID 12668495
- [Result] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Result] Yoshimoto D, Sakamoto Y, Uemura Y, Yamaguchi R, Naganawa H, Suzuki T. Comparative assessment of interatrial conduction delay during Bachmann's bundle pacing and right atrial appendage pacing using biatrial strain rate echocardiography. Heart Rhythm. 2025 Nov;22(11):2753-2754. doi: 10.1016/j.hrthm.2024.12.016. Epub 2024 Dec 15. No abstract available. PMID 39681277
- [Result] Bailin SJ, Adler S, Giudici M. Prevention of chronic atrial fibrillation by pacing in the region of Bachmann's bundle: results of a multicenter randomized trial. J Cardiovasc Electrophysiol. 2001 Aug;12(8):912-7. doi: 10.1046/j.1540-8167.2001.00912.x. PMID 11513442
- [Result] Johner N, Namdar M, Shah DC. Intra- and interatrial conduction abnormalities: hemodynamic and arrhythmic significance. J Interv Card Electrophysiol. 2018 Aug;52(3):293-302. doi: 10.1007/s10840-018-0413-4. Epub 2018 Aug 20. PMID 30128800
- [Result] Kawakami H, Ramkumar S, Nolan M, Wright L, Yang H, Negishi K, Marwick TH. Left Atrial Mechanical Dispersion Assessed by Strain Echocardiography as an Independent Predictor of New-Onset Atrial Fibrillation: A Case-Control Study. J Am Soc Echocardiogr. 2019 Oct;32(10):1268-1276.e3. doi: 10.1016/j.echo.2019.06.002. Epub 2019 Aug 26. PMID 31466848
- [Result] Infeld M, Habel N, Wahlberg K, Meagher S, Meyer M, Lustgarten D. Bachmann bundle potential during atrial lead placement: A case series. Heart Rhythm. 2022 Mar;19(3):490-494. doi: 10.1016/j.hrthm.2021.11.015. Epub 2021 Nov 12. No abstract available. PMID 34775070
- [Result] Zagoridis K, Koutalas E, Intzes S, Symeonidou M, Zagoridou N, Karagogos K, Spanoudakis E, Kanoupakis E, Kochiadakis G, Dinov B, Dagres N, Hindricks G, Bollmann A, Nedios S. P-wave duration and interatrial block as predictors of new-onset atrial fibrillation: A systematic review and meta-analysis. Hellenic J Cardiol. 2023 Jul-Aug;72:57-64. doi: 10.1016/j.hjc.2023.03.007. Epub 2023 Apr 5. PMID 37028490
- [Result] Vedage NA, Cronin EM. Effect of pacing site on P wave parameters: Within-patient comparison of right atrial appendage and Bachmann's bundle. J Electrocardiol. 2024 May-Jun;84:9-14. doi: 10.1016/j.jelectrocard.2024.02.006. Epub 2024 Feb 27. PMID 38432160
- [Result] Shali S, Su Y, Ge J. Interatrial septal pacing to suppress atrial fibrillation in patients with dual chamber pacemakers: A meta-analysis of randomized, controlled trials. Int J Cardiol. 2016 Sep 15;219:421-7. doi: 10.1016/j.ijcard.2016.06.093. Epub 2016 Jun 23. PMID 27371866
- [Result] Infeld M, Nicoli CD, Meagher S, Tompkins BJ, Wayne S, Irvine B, Betageri O, Habel N, Till S, Lobel J, Meyer M, Lustgarten DL. Clinical impact of Bachmann's bundle pacing defined by electrocardiographic criteria on atrial arrhythmia outcomes. Europace. 2022 Oct 13;24(9):1460-1468. doi: 10.1093/europace/euac029. PMID 35304608
- [Result] Lemery R, Guiraudon G, Veinot JP. Anatomic description of Bachmann's bundle and its relation to the atrial septum. Am J Cardiol. 2003 Jun 15;91(12):1482-5, A8. doi: 10.1016/s0002-9149(03)00405-3. No abstract available. PMID 12804741
- [Result] Kreimer F, Gotzmann M. Pacemaker-induced atrial fibrillation reconsidered-associations with different pacing sites and prevention approaches. Front Cardiovasc Med. 2024 Jun 18;11:1412283. doi: 10.3389/fcvm.2024.1412283. eCollection 2024. PMID 38957332
- [Result] Sweeney MO, Hellkamp AS, Ellenbogen KA, Greenspon AJ, Freedman RA, Lee KL, Lamas GA; MOde Selection Trial Investigators. Adverse effect of ventricular pacing on heart failure and atrial fibrillation among patients with normal baseline QRS duration in a clinical trial of pacemaker therapy for sinus node dysfunction. Circulation. 2003 Jun 17;107(23):2932-7. doi: 10.1161/01.CIR.0000072769.17295.B1. Epub 2003 Jun 2. PMID 12782566